CLINICAL TRIAL: NCT06515613
Title: A Phase 1, First in Human Study of CTIM-76, a Claudin-6 (CLDN6)-Directed Bispecific Antibody, in Patients With Recurring Ovarian Cancer and Other Advanced Solid Tumors
Brief Title: A Phase 1 Study of CTIM-76 in Patients With Recurring Ovarian Cancer and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-CTIM76-101
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Platinum-resistant Ovarian Cancer; Testicular Cancer; Endometrial Cancer
MeSH Terms: conditions — Testicular Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1a is a dose escalation assessing 9 different dose levels and phase 1b will evaluate 2 doses from the phase 1a.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTIM-76 (Experimental): Phase 1a: Dose Escalation-each dose cohort will assess toxicity 28 days following the first dose of CTIM76; anticipate a total of 9 dose cohorts.
  Phase 1b: Dose Expansion - 40 subjects will be evaluated using 2 different doses/dosing schedules of CTIM-76
  Interventions: Drug: CTIM-76

INTERVENTIONS:
Drug: CTIM-76 — CLDN6 bispecific Antibody administered weekly (Day 1, 8, 15 and 22) of a 28-day treatment cycle until disease progression.
  Other Names: CTIM-76 Claudin 6 bispecific Antibody

SUMMARY:
This is a Phase 1a/1b, open-label, dose escalation and expansion study to evaluate the safety and efficacy of CTIM-76 (study drug), a CLDN6-directed T cell-engaging bispecific antibody, in participants with platinum-refractory/resistant ovarian cancer (PRROC) and other advanced CLDN6-positive solid tumors (i.e., testicular and endometrial).

DETAILED DESCRIPTION:
The phase 1a Dose Escalation portion of the trial will enroll participants with PRROC, testicular, or endometrial cancer into one of approximately 9 dose escalation cohorts to assess safety, tolerability and to determine the recommended dose for expansion (RDE). CTIM-76 is to be administered once weekly (Q1W) for each cycle. A cycle is defined as 28 days. Participants will be dosed until documentation of disease progression, unacceptable toxicity, or participant/physician decision.

The phase 1b dose expansion phase will evaluate CTIM-76 in at least one indication at up to 2 doses and/or dosing schedules (n=20 response evaluable participants in each cohort ) in the dose expansion phase of the trial (Phase 1b) studying one of the following advanced solid tumor types: PROC, testicular, or endometrial. This is to enable dose- and exposure-response analyses. The expansion doses/dosing schedules for Phase 1b will be determined by Sponsor in conjunction with Safety Review Committee (SRC) based upon all available safety, pharmacokinetic (PK), pharmacodynamic (PD), biomarker and preliminary efficacy data from Phase 1a.

The selection of the RP2D will be based on the totality of data from Phase 1b.

ELIGIBILITY:
Inclusion Criteria:

* Participants with CLDN6 positive platinum resistant/refractory ovarian, advanced testicular or advanced endometrial cancer.
* Participants with measurable disease per RECIST 1.1.
* ECOG 0, 1, or 2 and life expectancy of ≥ 12 weeks.
* Participants with adequate organ function.

Exclusion Criteria:

* Evidence of central nervous system metastases, leptomeningeal disease or spinal cord compression.
* Uncontrolled significant active infection or any medical or other condition that in opinion of the Investigator would preclude the participant's participation in the study.
* Concurrent participation in another investigational clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | From date of first dose of CTIM-76 until 28 days following the first dose
  Phase 1a will evaluate increasing doses of CTIM-76 based on the assessment of DLTs
Overall response rate (ORR) | From date of first dose of CTIM-76 until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  ORR will be based on the best overall response rate as assessed by Investigators according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chagin, MD, Study Chair — Context Therapeutics Inc.
Locations (11):
- United States (11):
  - University of Arkansas Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - Precision NextGen Oncology & Research Center, Beverly Hills, California
  - SCRI at Denver Health, Denver, Colorado
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Providence Cancer Institute of Oregon, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - SCRI at Mary Crowley, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided